CLINICAL TRIAL: NCT03534570
Title: A Prospective Study on the Need of Gated (GAT) Radiotherapy in Left Sided Breast Cancer Patients Treated at the Technical University Munich (TUM) - the GATTUM Protocol
Brief Title: Gated Radiotherapy in Left Sided Breast Cancer Patients
Acronym: GATTUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Marciana Duma, M.D., Technical University of Munich
Other Study IDs: GATTUM -1
Record Dates: First submitted 2015-08-03; First posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Breast Neoplasm Female; Radiotherapy Side Effect; Heart Diseases
MeSH Terms: conditions — Radiation Injuries; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the need of respiratory gated radiotherapy in left sided breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* left sided breast cancer patients treated with breast conserving surgery

Exclusion Criteria:

* patients treated with mastectomy
* patients with positive lymph nodes

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: left sided breast cancer patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of distance from chestwall to the heart | 3 years
  Rigid and non-rigid measurement of distance from chestwall to the heart.
Measurement of distance from the heart to the mammary gland | 3 years
  Rigid and non-rigid measurement of distance from the heart to the mammary gland

CONTACTS AND LOCATIONS:
Overall Officials: Marciana Duma, M.D., Principal Investigator — Klinikum rechts der Isar, department of Radiation oncology
Locations (1):
- Klinikum rechts der Isar; TUM, Munich, Germany

REFERENCES:
- [Background] Fajardo LF, Stewart JR, Cohn KE. Morphology of radiation-induced heart disease. Arch Pathol. 1968 Nov;86(5):512-9. No abstract available. PMID 5681435
- [Background] Adams MJ, Lipsitz SR, Colan SD, Tarbell NJ, Treves ST, Diller L, Greenbaum N, Mauch P, Lipshultz SE. Cardiovascular status in long-term survivors of Hodgkin's disease treated with chest radiotherapy. J Clin Oncol. 2004 Aug 1;22(15):3139-48. doi: 10.1200/JCO.2004.09.109. PMID 15284266
- [Background] Shimizu Y, Kodama K, Nishi N, Kasagi F, Suyama A, Soda M, Grant EJ, Sugiyama H, Sakata R, Moriwaki H, Hayashi M, Konda M, Shore RE. Radiation exposure and circulatory disease risk: Hiroshima and Nagasaki atomic bomb survivor data, 1950-2003. BMJ. 2010 Jan 14;340:b5349. doi: 10.1136/bmj.b5349. PMID 20075151
- [Background] Andratschke N, Maurer J, Molls M, Trott KR. Late radiation-induced heart disease after radiotherapy. Clinical importance, radiobiological mechanisms and strategies of prevention. Radiother Oncol. 2011 Aug;100(2):160-6. doi: 10.1016/j.radonc.2010.08.010. Epub 2010 Sep 7. PMID 20826032
- [Background] Carmel RJ, Kaplan HS. Mantle irradiation in Hodgkin's disease. An analysis of technique, tumor eradication, and complications. Cancer. 1976 Jun;37(6):2813-25. doi: 10.1002/1097-0142(197606)37:63.0.co;2-s. PMID 949701
- [Background] Larsen RL, Jakacki RI, Vetter VL, Meadows AT, Silber JH, Barber G. Electrocardiographic changes and arrhythmias after cancer therapy in children and young adults. Am J Cardiol. 1992 Jul 1;70(1):73-7. doi: 10.1016/0002-9149(92)91393-i. PMID 1615874
- [Background] Cella L, Liuzzi R, Conson M, Torre G, Caterino M, De Rosa N, Picardi M, Camera L, Solla R, Farella A, Salvatore M, Pacelli R. Dosimetric predictors of asymptomatic heart valvular dysfunction following mediastinal irradiation for Hodgkin's lymphoma. Radiother Oncol. 2011 Nov;101(2):316-21. doi: 10.1016/j.radonc.2011.08.040. Epub 2011 Sep 16. PMID 21925755
- [Background] Duma MN, Molls M, Trott KR. From heart to heart for breast cancer patients - cardiovascular toxicities in breast cancer radiotherapy. Strahlenther Onkol. 2014 Jan;190(1):5-7. doi: 10.1007/s00066-013-0465-4. Epub 2013 Nov 21. No abstract available. PMID 24253182
- [Background] Darby SC, Ewertz M, McGale P, Bennet AM, Blom-Goldman U, Bronnum D, Correa C, Cutter D, Gagliardi G, Gigante B, Jensen MB, Nisbet A, Peto R, Rahimi K, Taylor C, Hall P. Risk of ischemic heart disease in women after radiotherapy for breast cancer. N Engl J Med. 2013 Mar 14;368(11):987-98. doi: 10.1056/NEJMoa1209825. PMID 23484825
- [Background] Bartlett FR, Colgan RM, Carr K, Donovan EM, McNair HA, Locke I, Evans PM, Haviland JS, Yarnold JR, Kirby AM. The UK HeartSpare Study: randomised evaluation of voluntary deep-inspiratory breath-hold in women undergoing breast radiotherapy. Radiother Oncol. 2013 Aug;108(2):242-7. doi: 10.1016/j.radonc.2013.04.021. Epub 2013 May 29. PMID 23726115
- [Background] Korreman SS, Pedersen AN, Josipovic M, Aarup LR, Juhler-Nottrup T, Specht L, Nystrom H. Cardiac and pulmonary complication probabilities for breast cancer patients after routine end-inspiration gated radiotherapy. Radiother Oncol. 2006 Aug;80(2):257-62. doi: 10.1016/j.radonc.2006.07.020. Epub 2006 Aug 14. PMID 16905210